CLINICAL TRIAL: NCT00691886
Title: Safety and Efficacy of Intravenous Dexmedetomidine Infusion During Flexible Bronchoscoy and Endobronchical Ultrasound
Brief Title: Safety and Efficacy of Intravenous (IV) Dexmedetomidine During Flexible Bronchoscopy and Endobronchial Ultrasound
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI left institution prior to enrollment
Sponsor: Lahey Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2008-011
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Pain
Keywords: sedation
MeSH Terms: conditions — Pain | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Subjects randomized to arm 1 of the study will recieve standard of care conscious sedation for EBUS; midasolam and or fentanyl.
- 2 (Active Comparator): Subjects undergoing EBUS randomized to arm 2 of the study will recieve demedetomadine hydrochloride plus standard of care conscious sedation
  Interventions: Drug: dexmedetomidine hydrochloride

INTERVENTIONS:
Drug: dexmedetomidine hydrochloride — Dose of 0.4ug/kg/hr to 1.5ug/kg/hr to achieve a RASS score of -1 to-3 during the bronchoscopy procedure. Dexmedetomidine will infused a half hour before the proceudure is started and will continue throughout the procedure. Traditional sedatives (midazolam and or fentanyl) will be given prn.
  Other Names: Precedex
  Arms: 2

SUMMARY:
To achieve safe,consistent, continuous sedation using Dexmedetomidine in advaced bronchoscopy procedures that may reduce the need for rapid pain sedative infusion.

DETAILED DESCRIPTION:
Dexmedetomidine hydrochloride as a single agent produces sedation, pain relief, anxiety redution, stable respiratory rates, and predictable cardiovascular responses. Dexmedetomidine facilitates patient comfort, compliance and comprehension by offering sedation with the ability to awaken patients. This study is being done to determine sedation efficacy and dosing; measure reduction or eliminate the need for rapid sedative infusion during bronchoscopy; improvement of patient comfort and safety during complex bronchoscopy; establish a new paradigm for moderate sedation during flexible bronchoscopy

ELIGIBILITY:
Inclusion Criteria:

* Adults between the age of 18 and 85
* Adults scheduled for flexible brochoscopy using EUBS (Endobronchial Ultrasound)

Exclusion Criteria:

* Sever bradycardia (rate < 50) and / or related bradydysrhymias (e.g. advanced heart block)
* Impaired ventricular functions (EF <30%)
* Hypovolemia or hypotension (SBP <90 or MAP <a55)
* Have GFR less than 15ml/min 1.73m2 or undergoing hemodialysis
* Endstage liver disease.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Achieve safe, consistent, continous moderate sedation using Dexmedetomidine in advanced bronchoscopy procedures, alleviating the need for rapid sedative infusion. | at conclusion of subject enrollemtn

CONTACTS AND LOCATIONS:
Overall Officials: David R Riker, MD, Principal Investigator — Lahey Clinic Medical Center
Locations (1):
- Lahey Clinic, Burlington, Massachusetts, United States